CLINICAL TRIAL: NCT07339748
Title: An Open-label, Multicenter Phase I/IIa Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ZL-85FA Tablets in Treating Advanced Solid Tumors
Brief Title: A Clinical Study of ZL-85FA Tablets
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ZL85-001
Record Dates: First submitted 2025-12-30; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Dose escalation group 1 (Experimental): ZL-85FA tablets 2.5mg
  Interventions: Drug: ZL-85FA tablets
- Dose escalation group 2 (Experimental): ZL-85FA tablets 5mg
  Interventions: Drug: ZL-85FA tablets
- Dose escalation group 3 (Experimental): ZL-85FA tablets 10mg
  Interventions: Drug: ZL-85FA tablets
- Dose escalation group 4 (Experimental): ZL-85FA tablets 15mg
  Interventions: Drug: ZL-85FA tablets
- Dose escalation group 5 (Experimental): ZL-85FA tablets 20mg
  Interventions: Drug: ZL-85FA tablets
- Dose escalation group 6 (Experimental): ZL-85FA tablets 25mg
  Interventions: Drug: ZL-85FA tablets
- Dose escalation group 7 (Experimental): ZL-85FA tablets 30mg
  Interventions: Drug: ZL-85FA tablets
- Dose extension group 1 (Experimental): Based on the results obtained from the dose escalation phase, the necessity and dosage of the IIa phase expansion cohort will be determined by the Drug Safety Review Committee (SMC) after discussion.
  Interventions: Drug: ZL-85FA tablets
- Dose extension group 2 (Experimental): Based on the results obtained from the dose escalation phase, the necessity and dosage of the IIa phase expansion cohort will be determined by the Drug Safety Review Committee (SMC) after discussion.
  Interventions: Drug: ZL-85FA tablets

INTERVENTIONS:
Drug: ZL-85FA tablets — ZL-85FA tablets 2.5mg, oral, once daily
  Arms: Dose escalation group 1
Drug: ZL-85FA tablets — ZL-85FA tablets 5mg, oral, once daily
  Arms: Dose escalation group 2
Drug: ZL-85FA tablets — ZL-85FA tablets 10mg, oral, once daily
  Arms: Dose escalation group 3
Drug: ZL-85FA tablets — ZL-85FA tablets 15mg, oral, once daily
  Arms: Dose escalation group 4
Drug: ZL-85FA tablets — ZL-85FA tablets 20mg, oral, once daily
  Arms: Dose escalation group 5
Drug: ZL-85FA tablets — ZL-85FA tablets 25mg, oral, once daily
  Arms: Dose escalation group 6
Drug: ZL-85FA tablets — ZL-85FA tablets 30mg, oral, once daily
  Arms: Dose escalation group 7
Drug: ZL-85FA tablets — Based on the results obtained from the dose escalation phase, the necessity and dosage of the IIa phase expansion cohort will be determined by the Drug Safety Review Committee (SMC) after discussion.
  Arms: Dose extension group 1
Drug: ZL-85FA tablets — Based on the results obtained from the dose escalation phase, the necessity and dosage of the IIa phase expansion cohort will be determined by the Drug Safety Review Committee (SMC) after discussion.
  Arms: Dose extension group 2

SUMMARY:
An open-label, multicenter phase I/IIa clinical study evaluating the safety, tolerability, pharmacokinetics, and preliminary efficacy of ZL-85FA tablets in treating advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

- 1.Voluntarily joining this study, signing informed consent form, good compliance, and able to cooperate with follow-up; 2.Age: >=18 years old and <=75 years old (including boundary values, calculated on the day of signing informed consent), gender not limited; 3.Patients with advanced breast cancer, ovarian cancer, fallopian tube cancer, primary peritoneal cancer, and prostate cancer confirmed by pathological histology or cytology.

4.ECOG <= 1 point; 5.Expected survival period >= 12 weeks; 6.Sufficient organ functio; 7. All acute toxicity reactions of previous anti-cancer treatments or surgical procedures have been relieved to baseline severity or NCI-CTCAE version 5.0 <= 1 (except for hair loss or other toxicity that the researcher considers to be of no safety risk to the patient); 8.Women and men of childbearing age should agree to take effective contraceptive measures (hormone or barrier therapy or abstinence) 10.During the study period and within 6 months after the end of the study; Female patients of childbearing age who have a negative serum or urine pregnancy test within 7 days before administration and must be non lactating patients.

Exclusion Criteria:

* 1.It is known that there is severe allergy to the investigational drug or any of its excipients (lactose, microcrystalline cellulose, low substituted hydroxypropyl cellulose, glyceryl behenate, hydroxypropyl methylcellulose, film coated premix (gastric soluble)); 2.Currently or previously suffering from other malignant tumors (excluding fully treated basal cell carcinoma or squamous cell carcinoma, cervical carcinoma in situ), unless curative treatment has been carried out and there is evidence of no recurrence or metastasis within the past 5 years; 3.Symptomatic central nervous system (CNS) metastases or asymptomatic CNS metastases requiring steroid treatment within 2 weeks prior to the first use of the study drug. Subjects with malignant meningitis or leptomeningeal spread; 4.Have received the last systemic anti-tumor treatment (chemotherapy, targeted therapy, immunotherapy, biologics, etc.) within 4 weeks before the first administration, with mitomycin or nitrosamines within 6 weeks, and small molecule targeted drugs within 2 weeks before the first administration of the study drug or within 5 half lives of the known drug (whichever is longer); Local palliative radiotherapy within 2 weeks prior to the first use of the study drug; The last administration of endocrine therapy is within 2 weeks before the first administration of the investigational drug (excluding necessary drug castration treatment for patients with metastatic castration resistant prostate cancer); Chinese herbal medicine or traditional Chinese patent medicines and simple preparations with anti-tumor indications were received within 2 weeks before the first administration of the study drug; 5.Individuals with severe infections within 4 weeks prior to the first administration, or those with active infections requiring oral or intravenous antibiotic treatment within 2 weeks prior; Individuals with active pulmonary tuberculosis who have undergone sufficient treatment before their first medication and have stopped anti tuberculosis treatment for at least 3 months are eligible for enrollment; 6.Receive blood transfusion, recombinant human thrombopoietin, recombinant human interleukin-11, erythropoietin, granulocyte colony-stimulating factor and other treatments within 2 weeks before the first use of the investigational drug; 7.Patients who have received systemic corticosteroid (prednisone>10 mg/day or equivalent doses of similar drugs, continuously used for more than 4 days) or other immunosuppressive therapy within 14 days before the first administration; Excluding the following situations: treatment with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids, and short-term prophylactic treatment with corticosteroids such as contrast agents.

  8.There are uncontrollable or significant cardiovascular and cerebrovascular diseases, including:
  1. Within 6 months prior to the first use of medication, there is a New York Heart Association (NYHA) grade II or higher congestive heart failure, unstable angina pectoris, myocardial infarction, or arrhythmia requiring treatment during screening, with a left ventricular ejection fraction (LVEF)<50%;
  2. Primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, and undifferentiated cardiomyopathy);
  3. Other cardiovascular and cerebrovascular diseases that have been determined by researchers to be unsuitable for inclusion.

  9.Uncontrollable electrolyte imbalances may affect the efficacy of QTc drugs , but retesting after intervention therapy is allowed; 10.Those who have undergone major surgeries requiring general anesthesia or have not withdrawn from other clinical trials within 4 weeks prior to the first administration; Within 2 weeks prior to enrollment, the patient has undergone surgery requiring local anesthesia/epidural anesthesia and has not yet recovered (excluding tissue biopsy); 11.he following active infections with clinical significance, including hepatitis B (HBV) and hepatitis C (HCV). Active hepatitis B is defined as: subjects who are HBsAg positive or HBcAb positive and whose HBV DNA is higher than the lower limit of detection (i.e. the upper limit of the normal value in the laboratory of each research center), if they reach the negative level of HBV DNA after antiviral treatment and receive antiviral drugs at least 2 weeks before the first administration, those who are willing to continue to receive anti hepatitis B virus treatment during the study period are allowed to be included in the study. Active hepatitis C is defined as those who are HCV antibody positive and whose HCV RNA is higher than the lower limit of detection (the upper limit of the normal value). Treponema pallidum antibody (TP Ab) positive and syphilis non-specific antibody titer (RPR) positive; 12.History of immunodeficiency, including positive human immunodeficiency virus (HIV) antibody test, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; 13.Patients with swallowing difficulties, chronic diarrhea, or oral absorption disorders; 14. Patients with bleeding tendency (for example, active peptic ulcer, recent hemorrhagic stroke [within 6 months before screening], proliferative diabetes retinopathy); 15.Within the first 4 weeks of enrollment, participated in other interventional clinical trials; 16.Other serious acute or chronic medical or psychiatric disorders or laboratory abnormalities that may increase the risk of participation in the study or increase the risk associated with the administration of the study drug, or interfere with the study results, as well as other situations where the researcher deems the patient unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate | Up to week 96
  defined as the proportion of subjects with an overall efficacy response of complete remission (CR) or partial remission (PR) after at least one post-baseline evaluation during the trial.

SECONDARY OUTCOMES:
Disease control rate | Up to week 96
  defined as the proportion of subjects with an overall efficacy response of CR, PR and stable disease (SD) after at least one post-baseline evaluation during the trial
Duration of response | Up to week 96
  defined as the duration from first remission (PR and CR) to disease progression or death
Progression free survival | Up to week 96
  defined as the time from first dose to disease progression or death
Overall survival | Up to week 96
  defined as the time from first dose to death

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No